CLINICAL TRIAL: NCT00124514
Title: Triptorelin for Ovary Protection in Childhood Onset Lupus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Watson Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Hermine Brunner, MD, Principal Investigator, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2008-1045; FD-R-00239 (Other Grant/Funding Number: FDA OOPD); NCT00088244 (obsolete NCT alias)
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Lupus; Ovarian damage; Menopause
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Triptorelin Pamoate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Triptorelin T1 (Experimental): Triptorelin Pamoate 25 μg/kg body weight
  Interventions: Drug: Triptorelin pamoate
- Triptorelin T2 (Experimental): Triptorelin Pamoate 50 μg/kg body weight
  Interventions: Drug: Triptorelin Pamoate
- Triptorelin T3 (Experimental): Triptorelin Pamoate 75 μg/kg body weight T3
  Interventions: Drug: Triptorelin Pamoate
- Triptorelin T4 (Experimental): Triptorelin Pamoate 100 μg/kg body weight T4
  Interventions: Drug: Triptorelin Pamoate
- Placebo (Placebo Comparator): Normal Saline
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Triptorelin pamoate — IM injection given monthly
  Other Names: Trelstar Depot
  Arms: Triptorelin T1
Drug: Triptorelin Pamoate — IM injection given monthly
  Other Names: Trelstar Depot
  Arms: Triptorelin T2
Drug: Triptorelin Pamoate — IM injection given monthly
  Other Names: Trelstar Depot
  Arms: Triptorelin T3
Drug: Triptorelin Pamoate — IM injection given monthly
  Other Names: Trelstar Depot
  Arms: Triptorelin T4
Other: placebo — placebo 0.9% normal saline IM injection
  Other Names: placebo 0.9% normal saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety of triptorelin when used for the protection of the ovaries (pair of female reproductive organs) during cyclophosphamide therapy for systemic lupus erythematosus (SLE; lupus) and to see what effects (good or bad) it has on patients. The study will be done with female patients who have been diagnosed with systemic lupus erythematosus, are younger than 21 years of age, and require intravenous cyclophosphamide to control the disease. Each patient will be in the study for approximately 23 months, until 4 months after the intravenous cyclophosphamide treatment has been completed.

This study is currently being conducted at 3 sites across the United States and Brazil (Los Angeles, Cincinnati and San Paulo Brazil). A total of 50 patients will participate in this study.

Each patient will be randomized (assigned) to one of 5 groups. Randomization means that patients are put into a group completely by chance. It is like flipping a coin. Neither the patient nor the study staff knows what group the patient is in. The patient has a 20% chance of being placed in any group.

This is a dose escalation study, each patient will receive the first dose of the study drug (T1 - T4, placebo). If a patient has complete ovarian suppression on day 27 after the initial injection of study drug, then she will remain on this weight-adjusted dose of study drug throughout the study. The dose will be increased up for a weight gain of 5kg or greater. The dose will not be adjusted downward for a weight loss. If COS was not maintained with the 1st dose of study drug, then the subsequently injected 2nd dose will be increased by 25% or at least 20 microgram/kg/dose. The maximal dose of 150 microgram/kg/dose will not be exceeded. The absolute maximum dose is 20 mg.

Funding Source: FDA OOPD and Watson Pharmaceuticals

DETAILED DESCRIPTION:
Lupus is an autoimmune disease that may harm all organs in the body and especially affects the kidney, brain, skin and lungs. Cyclophosphamide is a very effective medication to treat lupus, but it can damage the ovaries (pair of reproductive organs).

Only female lupus patients may participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Females under the age of 21 and non-pregnant
* Tanner stage of 2 or above as determined by physical examination of breast stage
* Diagnosis with SLE using the updated American College of Rheumatology (ACR) Classification Criteria for SLE 1
* Severe SLE requiring cyclophosphamide therapy
* Bone mineral density z-score > - 2.0
* Must be using a medically acceptable form of birth control during the study and must not be pregnant at the screening visit
* No clinically significant abnormal findings other than those consistent with the diagnosis of childhood-onset SLE (cSLE) on the physical examination, medical history or clinical laboratory results during screening
* Currently on any combination of medication but must not have been treated with more than one dose of cyclophosphamide or other gonadotoxic medications in the past
* Voluntary consent or, if under the age of consent, assent to participate in this study with permission by a legal guardian

Exclusion Criteria:

* Male patients of any age
* Female patients with a Tanner stage of 1
* Positive blood pregnancy test at screening or taking oral or injectable birth-control medications
* Prior exposure to more than one dose of gonadotoxic medications including cyclophosphamide
* History of allergic or adverse response to triptorelin
* Diagnosed with hypogonadism prior to cyclophosphamide exposure
* Acutely life-threatening disease activity that prohibits inclusion in a clinical trial
* History of clinically significant gastrointestinal tract, renal, hepatic, endocrine, oncologic, pulmonary (asthma accepted), or cardiovascular disease; or a history of tuberculosis, epilepsy, diabetes, depression, psychosis, or any other non-cSLE condition, which in the opinion of the physician, would jeopardize the safety of the subject or impact the validity of the study results
* Patient age 18 years of younger with severe depression as defined by a CDI (Children's Depression Inventory) score of > 23 or a patient age 19 to 21 years with severe depression as defined by a BDI (Beck's Depression Inventory) score > 29
* Patient admits to suicidal thoughts at screening visit
* Bone mineral density lower than z = -2.0.

Ages: 9 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2003-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hermine I Brunner, M.D. M.Sc., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (10):
- United States (9):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Memorial Hospital, Chicago, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morgan Stanley Children's Hospital of New York, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Hospital of Oklahoma, Oklahoma City, Oklahoma
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Brunner HI, Silva CA, Reiff A, Higgins GC, Imundo L, Williams CB, Wallace CA, Aikawa NE, Nelson S, Klein-Gitelman MS, Rose SR. Randomized, double-blind, dose-escalation trial of triptorelin for ovary protection in childhood-onset systemic lupus erythematosus. Arthritis Rheumatol. 2015 May;67(5):1377-85. doi: 10.1002/art.39024. PMID 25676588

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 130 patients were screened for the study and 31 were randomized to one of 5 arms to start. The arms determined the starting dose of Triptorelin. All arms participated in dose escalation until the subjects reached and maintained COS.
  2 subjects withdrew prior to start of study procedures.
Groups:
- Triptorelin T1: Triptorelin Pamoate 25 μg/kg body weight starting dose
  Dose escalation initiated if COS was not maintained with the 1st dose of study drug. The subsequently injected 2nd dose was increased by 25% or at least 20 μg/kg dose. This procedure of dose increases repeated until COS was maintained.
- Triptorelin T2: Triptorelin Pamoate 50 μg/kg body weight starting dose
  Dose escalation initiated if COS was not maintained with the 1st dose of study drug. The subsequently injected 2nd dose was increased by 25% or at least 20 μg/kg dose. This procedure of dose increases repeated until COS was maintained.
- Triptorelin T3: Triptorelin Pamoate 75 μg/kg body weight starting dose
  Dose escalation initiated if COS was not maintained with the 1st dose of study drug. The subsequently injected 2nd dose was increased by 25% or at least 20 μg/kg dose. This procedure of dose increases repeated until COS was maintained.
- Triptorelin T4: Triptorelin Pamoate 100 μg/kg body weight starting dose
  Dose escalation initiated if COS was not maintained with the 1st dose of study drug. The subsequently injected 2nd dose was increased by 25% or at least 20 μg/kg dose. This procedure of dose increases repeated until COS was maintained.
Period: Overall Study
Arm/Group | Placebo | Triptorelin T1 | Triptorelin T2 | Triptorelin T3 | Triptorelin T4
Started | 6 | 9 | 8 | 6 | 2
Completed | 2 | 7 | 7 | 5 | 1
Not Completed | 4 | 2 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Triptorelin T3: Triptorelin Pamoate 75 μg/kg body weight
- Triptorelin T4: Triptorelin Pamoate 100 μg/kg body weight
- Total: Total of all reporting groups
Arm/Group | Placebo | Triptorelin T1 | Triptorelin T2 | Triptorelin T3 | Triptorelin T4 | Total
Number analyzed (Participants) | 6 | 9 | 8 | 6 | 2 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.9 (2.1) | 15.9 (2.6) | 16.5 (2.2) | 13.0 (2.1) | 12.50 (0) | 15.4 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 8 | 6 | 2 | 31
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 4 | 4 | 2 | 15
  Not Hispanic or Latino | 2 | 8 | 4 | 2 | 0 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 0 | 2 | 1 | 9
  White | 5 | 3 | 6 | 4 | 1 | 19
  More than one race | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose of Triptorelin for Ovarian Suppression
Description: Dose escalation was initiated If COS was not maintained with the 1st dose of study drug. Subsequent doses were increased by 25% or at least 20μg/kg dose. This procedure of dose increases by 25% or at least 20μg/kg dose was repeated until COS was maintained. Absolute max dose 7.8mg. Triptorelin (T1-T4) groups were pooled for analysis.
Time Frame: baseline to week 24
Measure: Number; unit: μg/kg
Groups:
- Triptorelin (T1-T4): Due to the dose escalation during the study, Triptorelin (T1-T4) groups were pooled for analysis.
Arm/Group | Placebo | Triptorelin (T1-T4)
Number analyzed (Participants) | 4 | 21
μg/kg | NA — Ovarian suppression not reached in placebo group | 120

2. Secondary Outcome: Length of Time of Triptorelin Treatment to Achieve Ovarian Suppression
Description: Time to ovarian suppression, based on suppressed LH levels, after the initial dose of triptorelin. Due to the dose escalation during the study, Triptorelin (T1-T4) groups were pooled for analysis.
Time Frame: baseline to week 24
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Triptorelin: Triptorelin Pamoate
  Due to the dose escalation during the study, Triptorelin (T1-T4) groups were pooled for analysis.
Arm/Group | Placebo | Triptorelin
Number analyzed (Participants) | 4 | 21
days | NA [NA to NA] — Ovarian suppression not reached in placebo group | 18 [15 to 25]

ADVERSE EVENTS:
Description: Due to the dose escalation during the study, Triptorelin (T1-T4) groups were pooled for analysis.
Groups:
- Placebo Group: Normal Saline
  placebo: placebo 0.9% normal saline IM injection
Arm/Group | Placebo Group | Triptorelin
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/25
Serious Adverse Events (participants affected / at risk) | 3/6 | 4/25
Other Adverse Events (participants affected / at risk) | 3/6 | 6/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=6) | Triptorelin (N=25)
Oedema peripheral (General disorders) | 0 | 1 (2)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neuropsychiatric lupus (Nervous system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Diffuse vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=6) | Triptorelin (N=25)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Fatigue (General disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (4)
Hot flush (Vascular disorders) | 1 (1) | 5 (5)
Hypertension (Vascular disorders) | 0 (0) | 4 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Oedema (General disorders) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes